CLINICAL TRIAL: NCT01734356
Title: Molecular Mechanism Identification in Inherited Arrhythmias and Valvulopathies From Induced Pluripotent Stem Cells
Acronym: Diag-iPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Masking: None
Other Study IDs: BRD/10/11-P
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Inherited Arrhythmias and Valvulopathies
Keywords: iPS; fibroblast; arrhythmias; valvulopathies; electrophysiology; genetics
MeSH Terms: conditions — Arrhythmias, Cardiac

ARMS (3):
- inherited arrhythmias (Other): 6 patient with inherited arrhythmias
  Interventions: Other: Skin biopsies
- valvulopathies (Other): 6 patient with valvulopathies
  Interventions: Other: Skin biopsies
- controle (Other): 8 healthy people for these pathologies
  Interventions: Other: Skin biopsies

INTERVENTIONS:
Other: Skin biopsies

SUMMARY:
The recent developments of research on iPS (induced pluripotent stem) cells lead to the establishment of mature cell lines such as cardiomyocytes or valvular interstitial cells with genetic and cellular characteristics of the donors. These cells represent a biological material more readily available to identify the pathophysiological mechanisms involved in the diseases of BrS or ERS patients, which will lead to the identification of genetic markers.

ELIGIBILITY:
Inclusion criteria:

* Patient with a family history of inherited arrhythmia or valvulopathy
* Age : 22-60 yo.
* patient no confine to bed
* Male or female
* Written consent
* Patient affiliated to the French social security

Exclusion criteria:

* Pregnant woman
* Patient under 22 yo or adults under guardianship
* Indication against local anesthesia
* Anticoagulant treatment
* Absence or positivity of HIV, HBV, HCV serology

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Production of cardiomyocytes modele from skin fibroblast of arrhythmic patient

SECONDARY OUTCOMES:
Production of valve interstitial cells modele from skin fibroblast of patient with a valvulopathy

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PROBST, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France